CLINICAL TRIAL: NCT04228198
Title: Protocol of the Italian Radical Cystectomy Registry: a Non-randomized, 24-month, Multicenter Study Comparing Robotic-assisted, Laparoscopic, and Open Surgery for Radical Cystectomy in Bladder Cancer
Brief Title: Protocol of the Italian Radical Cystectomy Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Ettore De Berardinis, Researcher, University of Roma La Sapienza
Other Study IDs: R.I.C.
Record Dates: First submitted 2020-01-03; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radical cystectomy: Patients with histologically confirmed diagnosis of bladder cancer undergoing radical cystectomy surgery at 28 Urology departments in Italy
  Interventions: Procedure: Radical cystectomy

INTERVENTIONS:
Procedure: Radical cystectomy — Procedure/Surgery: Radical cystectomy. Removal of urinary bladder with three different approaches: i) Robotic-assisted, ii) Laparoscopic, and iii) Open Surgery

SUMMARY:
Background: Bladder cancer is the ninth most common type of cancer worldwide. In the past, Radical Cystectomy via open surgery has been considered the gold-standard treatment for muscle invasive bladder cancer. However, in recent years there has been a progressive increase in the use of robot-assisted laparoscopic radical cystectomy surgery. The aim of the current project is to investigate the surgical, oncological, and functional outcomes of patients with bladder cancer who undergo radical cystectomy surgery comparing three different surgical techniques (robotic-assisted, laparoscopic, and open surgery). Pre-, peri- and post-operative factors will be examined, and participants will be followed for a period of up to 24 months to identify risks of mortality, oncological outcomes, hospital readmission, sexual performance, and continence.

Methods: The study is an observational, prospective, multicenter, cohort study to assess patients affected by bladder neoplasms undergoing radical cystectomy and urinary diversion. The Italian Radical Cystectomy Registry is an electronic registry to prospectively collect the data of patients undergoing Radical Cystectomy conducted with any technique (open, laparoscopic, robotic-assisted). Twenty-eight urology departments across Italy will provide data for the study, with recruitment phase between 1st January 2017-31st June 2020). Information is collected from the patients at the moment of surgical intervention and during follow-up (3, 6, 12, and 24 months after radical cystectomy surgery). Peri-operative variables include surgery time, type of urinary diversion, conversion to open surgery, bleeding, nerves sparing and lymphadenectomy. Follow-up data collection includes histological information (e.g., post-op staging, grading and tumor histology), short- and long-term outcomes (e.g., mortality, post-op complications, hospital readmission, sexual potency, continence etc).

Discussion: The current protocol aims to contribute additional data to the field concerning the short- and long-term outcomes of three different radical cystectomy surgical techniques for patients with bladder cancer, including open, laparoscopic, and robot-assisted. This is a comparative-effectiveness trial that takes into account a complex range of factors and decision making by both physicians and patients that affect their choice of surgical technique.

DETAILED DESCRIPTION:
The aim of the project is to investigate the surgical, oncological, and functional outcomes of patients with bladder cancer who undergo radical cystectomy surgery comparing three different surgical techniques (robotic-assisted, laparoscopic, and open surgery). Pre-, peri- and post-operative factors will be examined, and participants will be followed for a period of up to 24 months to identify risks of mortality, oncological outcomes, hospital readmission, sexual performance, and continence.

Twenty-eight participating centers across Italy will provide data for the study: Urology Clinic, University of Bologna; Department of Urology, AOU Careggi, Florence; European Institute of Oncology Milan; San Raffaele Hospital, Milan; University Hospital of Verona; Department of Urology, Policlinico Abano; Department of Urology, Spedali Civili, Brescia; Department of Urology and Kidney Transplantation, University of Foggia, Foggia; Galliera Hospital, Genova; ASST Niguarda Metropolitan Hospital, Niguarda; Policlinico Umberto I, Saproma; Department of Clinical Urology, University of Perugia; Department of Clinical Urology, AOUP Cisanello Hospital, Pisa; Department of Clinical Urology, Palermo University, Palermo; Department of Clinical Urology, Alessandria Hospital, Alessandria; Department of Clinical Urology, ASST Mantova, Mantova; Department of Clinical Urology, ASL Abruzzo; Department of Clinical Urology Ca Foncello Hospital, Treviso; Department of Clinical Urology II, Bari University, Bari; Department of Clinical Urology, Vittorio Emanuele Hospital, Catania; Department of Clinical Urology, Casa Sollievo della Sofferenza, Sgrotondo; Hospital Bassiano, Bassano; Department of Clinical Urology, Hospital San Francesco ASL 3, Nuoro; Department of Clinical Urology, Portogruaro; Department of Clinical Urology, Biella Hospital, Biella; Department of Clinical Urology Chioggia Hospital; Ausl Modena; Department of Urology and Kidney Transplantation, Bianchi-Melacrino-Morelli Grand Metropolitan Hospital.

The inclusion criteria are: 1) male and female consecutively recruited patients; 2) age ≥18 years; 3) histologically confirmed diagnosis of bladder cancer eligible for radical cystectomy surgery at date of enrollment; 4) providing written, informed consent.

At baseline and after 3, 6, 12, and 24 months post-surgery, data will be taken directly from the patients at their follow-up medical visits and entered into the online database. The physician identifying and recruiting patients is in charge of completing the data collection forms during follow-up, even if the patient is subsequently treated in another center.

Variables of interest include demographic variables (age, sex, etc), surgical factors (technique use, length of surgery, blood loss, type of urinary diversion, node burden, histological exams, surgical margins etc), mortality, morbidity (pre-, during- and post-surgery), oncological results, and functioning (continence and sexual performance) over follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male and female consecutively recruited patients
* Age ≥18 years
* Histologically confirmed diagnosis of bladder cancer eligible for radical cystectomy surgery (according to EAU guidelines) at date of enrollment
* Providing written, informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population is composed of subjects affected by bladder cancer that will undergo radical cystectomy. Surgery has been than divided in three different approaches: laparoscopic, robot-assisted and open.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Surgery time | Baseline
  Total surgery time, in minutes during surgery at baseline
Type of urinary diversion | Baseline
  Type of urinary diversion performed during the cystectomy surgery at baseline
Eventual conversion to open surgery | Baseline
  If the surgery technique changes from laproscopic surgery to open surgery during the intervention at baseline
Amount of surgical blood loss | Baseline
  Amount of blood lost during the surgical procedure at baseline in milliliters
Number of participants who underwent nerve-sparing | Baseline
  Nerve sparing during baseline surgery (no/unilateral/bilateral)
Number of participants who underwent lymphadenectomy | Baseline
  lymphadenectomy (not performed/ bilateral external iliac nodes /bilateral presacral iliac) during baseline surgery

SECONDARY OUTCOMES:
Histological evaluation of all patients | Immediately after surgery
  Tumor histology, (transitional cell carcinoma, adenocarcinoma, or other)
Rate of Mortality | Up to 24 months
  All-cause mortality after surgery
Rate of Hospitalization | Up to 24 months
  Any in-patient hospitalization in teh 24 months following surgical discharge.
Sexual potency rates | Up to 24 months
  Sexual potency in the patient following surgery. Self-reported.
Continence rates | Up to 24 months
  Daytime and nighttime continence following surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- policlinico Umberto I - Department of Gynecological-Obstetrics Sciences and Urological Sciences, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Porreca A, Palmer K, Artibani W, Antonelli A, Bianchi L, Brunocilla E, Bocciardi AM, Brausi M, Busetto GM, Carini M, Carrieri G, Celia A, Cindolo L, Cochetti G, Colombo R, De Berardinis E, De Cobelli O, Di Maida F, Ercolino A, Gaboardi F, Galfano A, Gallina A, Gallucci M, Introini C, Mearini E, Minervini A, Montorsi F, Musi G, Pini G, Schiavina R, Secco S, Serni S, Simeone C, Tasso G, D'Agostino D. Protocol of the Italian Radical Cystectomy Registry (RIC): a non-randomized, 24-month, multicenter study comparing robotic-assisted, laparoscopic, and open surgery for radical cystectomy in bladder cancer. BMC Cancer. 2021 Jan 11;21(1):51. doi: 10.1186/s12885-020-07748-7. PMID 33430820